CLINICAL TRIAL: NCT04021043
Title: Phase I/II Trial of Ipilimumab or Nivolumab With BMS-986156 and Hypofractionated Stereotactic Radiation Therapy in Patients With Advanced Solid Malignancies
Brief Title: BMS-986156, Ipilimumab, and Nivolumab With or Without Stereotactic Body Radiation Therapy in Treating Patients With Advanced or Metastatic Lung/Chest or Liver Cancers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0419; NCI-2019-00405 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0419 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-02-01; First posted 2019-07-16 (Actual); Results first posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Advanced Malignant Solid Neoplasm; Metastatic Carcinoma in the Liver; Metastatic Carcinoma in the Lung; Metastatic Malignant Neoplasm in the Thoracic Cavity; Metastatic Malignant Solid Neoplasm
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Ipilimumab; CTLA-4 Antigen; Nivolumab; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group I (ipilimumab, BMS-986156, nivolumab) (Experimental): Patients receive ipilimumab IV over 90 minutes and anti-GITR agonistic monoclonal antibody BMS-986156 IV over 60 minutes on day 1. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Beginning day 1 of cycle 5 (day 85), patients receive nivolumab IV over 30 minutes. Treatment repeats every 28 days for up to 26 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Anti-GITR Agonistic Monoclonal Antibody BMS-986156; Biological: Ipilimumab; Biological: Nivolumab
- Group II (ipilimumab, BMS-986156, SBRT, nivolumab) (Experimental): Patients receive ipilimumab IV over 90 minutes and anti-GITR agonistic monoclonal antibody BMS-986156 IV over 60 minutes on day 1. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. After completion of cycle 2, patients then undergo SBRT on days 29-32 for 4 fractions or on days 29-40 for 10 fractions. Beginning day 1 of cycle 5 (day 85), patents receive nivolumab IV over 30 minutes. Treatment repeats every 28 days for up to 26 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Anti-GITR Agonistic Monoclonal Antibody BMS-986156; Biological: Ipilimumab; Biological: Nivolumab; Radiation: Stereotactic Body Radiation Therapy
- Group III (nivolumab, BMS-986156, SBRT) (Experimental): Patients receive nivolumab IV over 30 minutes and anti-GITR agonistic monoclonal antibody BMS-986156 over 60 minutes on day 1. Patients also undergo SBRT over 30-45 minutes on days 1-4 for 4 fractions or on days 1-12 for 10 fractions. Treatment repeats every 28 days for up to 26 cycles of nivolumab and for up to 4 cycles of anti-GITR agonistic monoclonal antibody BMS-986156 in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Anti-GITR Agonistic Monoclonal Antibody BMS-986156; Biological: Nivolumab; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Drug: Anti-GITR Agonistic Monoclonal Antibody BMS-986156 — Given IV
  Other Names: Anti-GITR MoAb BMS-986156; BMS 986156; BMS-986156; GITR Agonist BMS-986156; TNFRSF18 Agonist BMS-986156
Biological: Ipilimumab — Given IV
  Other Names: Anti-Cytotoxic T-Lymphocyte-Associated Antigen-4 Monoclonal Antibody; BMS-734016; MDX-010; MDX-CTLA4; Yervoy
  Arms: Group I (ipilimumab, BMS-986156, nivolumab); Group II (ipilimumab, BMS-986156, SBRT, nivolumab)
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation Therapy
  Arms: Group II (ipilimumab, BMS-986156, SBRT, nivolumab); Group III (nivolumab, BMS-986156, SBRT)

SUMMARY:
This phase I/II trial studies the side effects and best dose of anti-glucocorticoid-induced tumor necrosis factor receptor (GITR) agonistic monoclonal antibody BMS-986156 (BMS-986156) when given together with ipilimumab and nivolumab with or without stereotactic body radiation therapy and to see how well they work in treating patients with lung/chest or liver cancer that has spread to other places in the body. Immunotherapy with monoclonal antibodies, such as BMS-986156, ipilimumab, and nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Stereotactic body radiation therapy uses special equipment to position a patient and deliver radiation to tumors with high precision. This method can kill tumor cells with fewer doses over a shorter period and cause less damage to normal tissue. It is not yet known whether giving BMS-986156, ipilimumab, and nivolumab with or without stereotactic body radiation therapy will work better in treating patients with lung/chest or liver cancers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safe dose of BMS-986156 and dose limiting toxicities (DLT) (30 mg versus [vs] 100 mg) when combined with ipilimumab (3 mg/kg) for patients with metastatic cancer.

II. To evaluate the safety and toxicity profile of ipilimumab (3mg/kg) with BMS-986156 (30 or 100 mg) administered in combination with stereotactic body radiation therapy (SBRT) targeting 1-4 LIVER lesion(s) for patients with metastatic cancers.

III. To evaluate the safety and toxicity profile of ipilimumab (3mg/kg) with BMS-986156 (30 or 100 mg) administered in combination with SBRT targeting 1-4 LUNG lesion(s) for patients with metastatic cancer.

IV. To determine safety and toxicity profile of nivolumab (480 mg) with BMS-986156 (30 mg) administered in combination with SBRT targeting 1-4 LIVER lesion(s) for patients with metastatic cancers.

V. To determine safety and toxicity profile of nivolumab (480 mg) with BMS-986156 (30 mg) administered in combination with SBRT targeting 1-4 LUNG lesion(s) for patients with metastatic cancers.

SECONDARY OBJECTIVES:

I. To determine antitumor activity of ipilimumab therapy with BMS-986156 (30 or 100 mg) as well as nivolumab with BMS-986156 (30 mg) with SBRT treatment for 1-4 lung lesions in both the SBRT treated lesion and non-irradiate tumors.

II. To determine antitumor activity of ipilimumab therapy with or without BMS-986156 (30 or 100 mg) as well as nivolumab with BMS-986156 (30 mg) with SBRT treatment for 1-4 liver lesions in both the SBRT treated lesion and non-irradiate tumors.

III. To compare response and progression of the non-irradiated tumors between BMS-986156 with ipilimumab vs BMS-986156 with nivolumab, using both immune-related response criteria (irRC) and Response Evaluation Criteria in Solid Tumors (RECIST) version (V) 1.1.

IV. To evaluate the predictive potential value of tumor-associated and systemic immune biomarkers for therapy effectiveness and toxicity prediction.

V. To evaluate whether skeletal mass, neutrophil, neutrophil to lymphocyte ratio, and tumor bulk are correlated with clinical outcomes and adverse events.

VI. To evaluate whether tumor kinetics in combination with clinical correlates can help determine treatment response.

VII. To evaluate whether tumor mutational burden correlates with improved clinical outcomes and response criteria.

OUTLINE: This is a phase I, dose-escalation study of anti-GITR agonistic monoclonal antibody BMS-986156, followed by a phase II study. Patients are assigned to 1 of 3 groups.

GROUP I: Patients receive ipilimumab intravenously (IV) over 90 minutes and anti-GITR agonistic monoclonal antibody BMS-986156 IV over 60 minutes on day 1. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Beginning day 1 of cycle 5 (day 85), patients receive nivolumab IV over 30 minutes. Treatment repeats every 28 days for up to 26 cycles in the absence of disease progression or unacceptable toxicity.

GROUP II: Patients receive ipilimumab IV over 90 minutes and anti-GITR agonistic monoclonal antibody BMS-986156 IV over 60 minutes on day 1. Treatment repeats every 21 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. After completion of cycle 2, patients then undergo SBRT on days 29-32 for 4 fractions or on days 29-40 for 10 fractions. Beginning day 1 of cycle 5 (day 85), patents receive nivolumab IV over 30 minutes. Treatment repeats every 28 days for up to 26 cycles in the absence of disease progression or unacceptable toxicity.

GROUP III: Patients receive nivolumab IV over 30 minutes and anti-GITR agonistic monoclonal antibody BMS-986156 over 60 minutes on day 1. Patients also undergo SBRT over 30-45 minutes on days 1-4 for 4 fractions or on days 1-12 for 10 fractions. Treatment repeats every 28 days for up to 26 cycles of nivolumab and for up to 4 cycles of anti-GITR agonistic monoclonal antibody BMS-986156 in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days, then every 2-4 months for up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histological confirmation of solid metastatic cancer with at least one metastatic or primary lesion in the liver or lung/chest, except for group 1.
* Patients who have completed prior systemic anti-cancer therapies, an interval of 5 drug half-lives or 4-weeks whichever is shorter, is required, prior to enrollment on study. Note: patients with anaplastic thyroid will be waived from this inclusion criteria given the rapid trajectory of their disease
* All patients must have at least one metastatic or primary lesion within the lung/chest or liver located in an anatomical location amenable to SBRT treatment with 50 Gy in 4 fractions or with 60 Gy in 10 fractions, except for group 1.
* Repeat radiation in fields previously radiated will be allowed at the discretion of the treating physician
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky > 60%)
* Total bilirubin =< 2.0 mg/dL (does NOT apply to patients with Gilbert's syndrome) (use of growth factors or blood transfusion to achieve these requirements is not allowed 2 weeks prior to study enrollment)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) < 2.5 x institutional upper limit of normal (use of growth factors or blood transfusion to achieve these requirements is not allowed 2 weeks prior to study enrollment)
* White blood count (WBC) >= 2500/uL (use of growth factors or blood transfusion to achieve these requirements is not allowed 2 weeks prior to study enrollment)
* Absolute neutrophil count (ANC) >= 1000/uL (use of growth factors or blood transfusion to achieve these requirements is not allowed 2 weeks prior to study enrollment)
* Platelets >= 75K (use of growth factors or blood transfusion to achieve these requirements is not allowed 2 weeks prior to study enrollment)
* Hemoglobin >= 9 g/dL (use of growth factors or blood transfusion to achieve these requirements is not allowed 2 weeks prior to study enrollment)
* Creatinine =< 2.0 x upper limit of normal (ULN) (use of growth factors or blood transfusion to achieve these requirements is not allowed 2 weeks prior to study enrollment)
* Patients must be willing and able to review, understand, and provide written consent before starting therapy
* Patients with brain metastasis will be included as long as they are free of neurologic symptoms related to metastatic brain lesions and who do not require or receive systemic corticosteroid therapy, > 10 mg/day in the 14 days prior to beginning the trial (=< 10 mg steroid, e.g.: prednisone, is allowed). Patients with stable brain metastases (clinically and radiographically) for >= 4 weeks to enroll on the protocol.
* Patients that have previously progressed on immunotherapy such as ipilimumab, anti-PD-I, anti-PDL-1 or talimogene laherparepvec (T-VEC) will be eligible.

Exclusion Criteria:

* Serious autoimmune disease at the discretion of the treating attending: patients with a history of active serious inflammatory bowel disease (including Crohn's disease and ulcerative colitis) and autoimmune disorders such as rheumatoid arthritis, systemic progressive sclerosis (scleroderma), systemic lupus erythematosus or autoimmune vasculitis (e.g., Wegener's granulomatosis) are excluded from this study
* Active diverticulitis, intra-abdominal abscess, gastrointestinal (GI) obstruction, abdominal carcinomatosis or other known risk factors for bowel perforation
* Any underlying medical or psychiatric condition, which in the opinion of the Investigator, will make the administration of study drug hazardous or obscure the interpretation of adverse events (AEs): e.g. a condition associated with frequent diarrhea or chronic skin conditions, recent surgery or colonic biopsy from which the patient has not recovered, or partial endocrine organ deficiencies
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, history of congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Known active human immunodeficiency virus (HIV), hepatitis B, or hepatitis C that has not been documented to be stable
* Any non-oncology vaccine therapy used for prevention of infectious diseases (for up to one month prior to or after any dose of ipilimumab)
* Concomitant therapy with any of the following: IL-2, interferon or other non-study immunotherapy regimens; cytotoxic chemotherapy; immunosuppressive agents; other investigational therapies; or chronic use of systemic corticosteroids while receiving ipilimumab (as long as steroid replacement is significantly greater than what is required for physiologic replacement, i.e. in hypothyroidism)
* Pregnant women are excluded from this study. Women of child-bearing potential (WOCBP) must have a pregnancy test every 4 weeks and WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) within 24 hours prior to the start of immunotherapy drugs (ipilimumab/nivolumab/BMS-986156), during the course of the treatment and 160 days AFTER the last dose of study drug you should not get pregnant or breast feed. In the case of male participants, during the course of treatment and 220 days AFTER the last dose of immunotherapy you should not father a child (condom use is mandatory, even if vasectomized) or donate sperm. For contraception guidelines please see protocol
* History of or current immunodeficiency disease or prior treatment compromising immune function at the discretion of the treating physician
* Prior allogeneic stem cell transplantation
* Patients who were intolerant to previous immuno-oncology (IO) drugs should be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2019-08-19 (Actual); Primary Completion 2025-04-14 (Actual); Study Completion 2025-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joe Chang, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Chang JY, Xu X, Shroff GS, Comeaux NI, Li W, Rodon Ahnert J, Karp DD, Dumbrava EE, Verma V, Chen A, Welsh J, Hong DS. Phase I/II study of BMS-986156 with ipilimumab or nivolumab with or without stereotactic ablative radiotherapy in patients with advanced solid malignancies. J Immunother Cancer. 2024 Oct 9;12(10):e009975. doi: 10.1136/jitc-2024-009975. PMID 39384194
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment period: 08/2019 to 12/2021; Location: Single center trial that recruited patients at one hospital site (MD Anderson Cancer Center, Houston, TX)
Pre-assignment Details: Three patients on theIpilimumab + BMS-986156 (30 mg/kg) arm, one patient on Ipilimumab + BMS-986156 (100 mg/kg) arm and one patient on the Ipilimumab + BMS-986156 with SBRT arm discontinued BMS-986156 with Ipilimumab due to treatment-related adverse events.
Groups:
- Ipilimumab + BMS-986156 (30 mg/kg) Arm: Group 1: Administered four cycles of Ipilimumab (3 mg/kg) + BMS-986156 (30 mg as dose level 1) every 3 weeks.
- Ipilimumab + BMS-986156 (100 mg/kg) Arm: Group 1: Administered four cycles of Ipilimumab (3 mg/kg) + BMS-986156 (100 mg as dose level 2) every 3 weeks.
- Ipilimumab + BMS-986156 With SBRT Arm: Group 2: Administered four cycles of Ipilimumab (3 mg/kg) + BMS-986156 (100 mg) every 3 weeks with SABR (50 Gy/4 fx or 60-70 Gy/10 fx to liver/lung lesions).
- Nivolumab + BMS-986156 With SBRT Arm: Group 3: Administered four cycles of nivolumab (480 mg) + BMS-986156 (30 mg), every 4 weeks with SABR. Maintenance nivolumab given up to 2 years.
Period: Overall Study
Arm/Group | Ipilimumab + BMS-986156 (30 mg/kg) Arm | Ipilimumab + BMS-986156 (100 mg/kg) Arm | Ipilimumab + BMS-986156 With SBRT Arm | Nivolumab + BMS-986156 With SBRT Arm
Started | 10 | 10 | 10 | 20
Completed | 0 | 0 | 0 | 1
Not Completed | 10 | 10 | 10 | 19
Not completed — Adverse Event | 3 | 1 | 1 | 0
Not completed — Death | 2 | 3 | 1 | 3
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 6
Not completed — Discontinued due to disease progression | 4 | 5 | 7 | 10

BASELINE CHARACTERISTICS:
Groups:
- Ipilimumab + BMS-986156 Arm (30 mg/kg): Group 1: Administered four cycles of Ipilimumab (3 mg/kg) + BMS-986156 (30 mg as dose level 1) every 3 weeks.
- Ipilimumab + BMS-986156 Arm (100 mg/kg): Group 1: Administered four cycles of Ipilimumab (3 mg/kg) + BMS-986156 (100 mg as dose level 2) every 3 weeks.
- Total: Total of all reporting groups
Arm/Group | Ipilimumab + BMS-986156 Arm (30 mg/kg) | Ipilimumab + BMS-986156 Arm (100 mg/kg) | Ipilimumab + BMS-986156 With SBRT Arm | Nivolumab + BMS-986156 With SBRT Arm | Total
Number analyzed (Participants) | 10 | 10 | 10 | 20 | 50
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 59 [51 to 71] | 61 [49 to 77] | 65 [52 to 70] | 60 [52 to 68] | 61 [52 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 4 | 5 | 20
  Male | 4 | 5 | 6 | 15 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 0 | 1 | 3
  Not Hispanic or Latino | 8 | 10 | 10 | 19 | 47
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 1 | 3
  White | 7 | 10 | 9 | 18 | 44
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 0 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 10 | 20 | 50

OUTCOME MEASURES:

1. Primary Outcome: Number of Dose Limiting Toxicities (DLTs)
Description: Evaluate dose of BMS-986156 (30 mg vs 100 mg) and dose limiting toxicities (DLTs) when combined with ipilimumab (3 mg/kg), and evaluate DLTs when BMS-986156 administered in combination with ipilimumab (3 mg/kg) or nivolumab (480 mg) with SABR
Time Frame: Median duration of follow-up 32.3 months (95% CI 8.6 to 56.0)
Measure: Number; unit: Dose limiting toxicities
Arm/Group | Ipilimumab + BMS-986156 Arm (30 mg/kg) | Ipilimumab + BMS-986156 Arm (100 mg/kg) | Ipilimumab + BMS-986156 With SBRT Arm | Nivolumab + BMS-986156 With SBRT Arm
Number analyzed (Participants) | 10 | 10 | 10 | 20
Dose limiting toxicities | 1 | 1 | 0 | 0

2. Secondary Outcome: Assess SBRT and Palliative Radiation Completion
Description: Explore antitumor activity with SBRT and palliative radiation.
Time Frame: Median duration of follow-up 32.3 months (95% CI 8.6 to 56.0)
Population: Patients in the Ipilimumab + BMS-986156 Arm were not treated with SBRT and were not assessed for this Outcome Measure
Measure: Number; unit: Count of participants
Arm/Group | Ipilimumab + BMS-986156 Arm (30 mg/kg) | Ipilimumab + BMS-986156 Arm (100 mg/kg) | Ipilimumab + BMS-986156 With SBRT Arm | Nivolumab + BMS-986156 With SBRT Arm
Number analyzed (Participants) | 0 | 0 | 10 | 20
Count of participants
  Completion of SBRT without interruption due to RT-related AEs |  |  | 10 | 20
  Re-induction of SBRT due to progression per protocol |  |  | 0 | 4
  Received palliative RT while receiving immunotherapy |  |  | 0 | 3
  Received palliative RT after finishing all protocol-specified therapy |  |  | 2 | 5

3. Secondary Outcome: Immune-related Tumor Response
Description: Number of immune related responses of different immunotherapy schemes with or without SABR; Assessing complete response (CR), partial response (PR), and stable disease (SD)
Time Frame: Median duration of follow-up 32.3 months (95% CI 8.6 to 56.0)
Measure: Number; unit: Count of participants
Arm/Group | Ipilimumab + BMS-986156 Arm (30 mg/kg) | Ipilimumab + BMS-986156 Arm (100 mg/kg) | Ipilimumab + BMS-986156 With SBRT Arm | Nivolumab + BMS-986156 With SBRT Arm
Number analyzed (Participants) | 10 | 10 | 10 | 20
Count of participants
  Immune Related Stable Disease (irSD) | 2 | 1 | 4 | 7
  Immune Related Partial Response (irPR) | 1 | 0 | 0 | 2
  Immune Related Progressive Disease (irPD) | 1 | 5 | 5 | 14

4. Secondary Outcome: Out-of-field (Abscopal) Disease Control Rate (ACR)
Description: Patient's change of tumor since intiation of treatment and patient's exhibiting out of field disease control.
Time Frame: Median duration of follow-up 32.3 months (95% CI 8.6 to 56.0)
Population: Patients in the Ipilimumab + BMS-986156 Arms were not treated with SBRT and were not assessed for this Outcome Measure
Measure: Number; unit: Count of participants
Arm/Group | Ipilimumab + BMS-986156 Arm (30 mg/kg) | Ipilimumab + BMS-986156 Arm (100 mg/kg) | Ipilimumab + BMS-986156 With SBRT Arm | Nivolumab + BMS-986156 With SBRT Arm
Number analyzed (Participants) | 0 | 0 | 10 | 20
Count of participants
  Abscopal control rate |  |  | 7 | 9
  Disease control rate |  |  | 1 | 7

5. Secondary Outcome: Out-of-field (Abscopal) Response Rate (ARR)
Description: Assesses partial response (PR) rate and complete response (CR) rate
Time Frame: Median duration of follow-up 32.3 months (95% CI 8.6 to 56.0)
Measure: Number; unit: Count of participants
Arm/Group | Ipilimumab + BMS-986156 Arm (30 mg/kg) | Ipilimumab + BMS-986156 Arm (100 mg/kg) | Ipilimumab + BMS-986156 With SBRT Arm | Nivolumab + BMS-986156 With SBRT Arm
Number analyzed (Participants) | 10 | 10 | 10 | 20
Count of participants
  Objective Response Rate (ORR) | 1 | 0 | 0 | 2
  Abscopal response rate (ARR) | NA — Patients not treated with SBRT on this arm | NA — Patients not treated with SBRT on this arm | 0 | 2

6. Secondary Outcome: Tumor Burden: Disease Control Rate
Description: Assessing complete response (CR), partial response (PR), and stable disease (SD)
Time Frame: Median duration of follow-up 32.3 months (95% CI 8.6 to 56.0)
Measure: Number; unit: Count of participants
Arm/Group | Ipilimumab + BMS-986156 Arm (30 mg/kg) | Ipilimumab + BMS-986156 Arm (100 mg/kg) | Ipilimumab + BMS-986156 With SBRT Arm | Nivolumab + BMS-986156 With SBRT Arm
Number analyzed (Participants) | 10 | 10 | 10 | 20
Count of participants | 3 | 3 | 4 | 11

ADVERSE EVENTS:
Time Frame: Baseline to at least 100 days after the last dose of study treatment, up to 5 years.
Arm/Group | Ipilimumab + BMS-986156 Arm (30 mg/kg) | Ipilimumab + BMS-986156 Arm (100 mg/kg) | Ipilimumab + BMS-986156 With SBRT Arm | Nivolumab + BMS-986156 With SBRT Arm
All-Cause Mortality (participants affected / at risk) | 2/10 | 3/10 | 1/10 | 3/20
Serious Adverse Events (participants affected / at risk) | 6/10 | 10/10 | 5/10 | 9/20
Other Adverse Events (participants affected / at risk) | 10/10 | 10/10 | 10/10 | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ipilimumab + BMS-986156 Arm (30 mg/kg) (N=10) | Ipilimumab + BMS-986156 Arm (100 mg/kg) (N=10) | Ipilimumab + BMS-986156 With SBRT Arm (N=10) | Nivolumab + BMS-986156 With SBRT Arm (N=20)
Colitis (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 2
Diarrhea (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0
Hepatobiliary disorders - Other, specify (Gastrointestinal disorders) | 0 | 0 | 2 | 2
Thromboembolic event (Vascular disorders) | 2 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0
Hypercalcemia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pelvic pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Delirium (Nervous system disorders) | 1 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 1 | 0 | 0
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Anorectal infection (Infections and infestations) | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Cardiac disorders - Other, specify (Cardiac disorders) | 0 | 0 | 1 | 1
Dehydration (General disorders) | 1 | 0 | 0 | 0
Dysphagia (General disorders) | 0 | 0 | 1 | 1
Gastric hemorrhage (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Headache (General disorders) | 0 | 0 | 1 | 1
Hypoxia (General disorders) | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 1
Penile pain (General disorders) | 0 | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1 | 1
Spermatic cord obstruction (General disorders) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Vasovagal reaction (Nervous system disorders) | 0 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Blood bilirubin increased (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Death NOS (General disorders) | 5 | 1 | 3 | 3
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify * (General disorders) | 3 | 2 | 1 | 1
Encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ipilimumab + BMS-986156 Arm (30 mg/kg) (N=10) | Ipilimumab + BMS-986156 Arm (100 mg/kg) (N=10) | Ipilimumab + BMS-986156 With SBRT Arm (N=10) | Nivolumab + BMS-986156 With SBRT Arm (N=20)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7 | 2 | 10 | 10
Fatigue (General disorders) | 7 | 2 | 7 | 7
Abdominal pain (General disorders) | 6 | 2 | 7 | 7
Anorexia (General disorders) | 5 | 3 | 6 | 6
Back pain (General disorders) | 5 | 0 | 9 | 9
Rash (Skin and subcutaneous tissue disorders) | 8 | 1 | 4 | 4
Diarrhea (Gastrointestinal disorders) | 6 | 3 | 3 | 3
Aspartate aminotransferase increased (Gastrointestinal disorders) | 4 | 5 | 3 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 4 | 4
Edema limbs (Blood and lymphatic system disorders) | 5 | 0 | 5 | 5
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 6 | 0 | 4 | 4
Nausea (Gastrointestinal disorders) | 5 | 2 | 3 | 3
Chest wall pain (General disorders) | 0 | 2 | 7 | 7
Creatinine increased (Renal and urinary disorders) | 4 | 2 | 3 | 3
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 2 | 4 | 3 | 3
Weight loss (Metabolism and nutrition disorders) | 5 | 1 | 3 | 3
Anemia (Blood and lymphatic system disorders) | 4 | 2 | 4 | 4
Fever (General disorders) | 4 | 0 | 4 | 4
General disorders and administration site conditions - Other, specify (General disorders) | 5 | 3 | 0 | 0
Pain (General disorders) | 3 | 1 | 4 | 4
Alanine aminotransferase increased (Gastrointestinal disorders) | 5 | 3 | 2 | 2
Hypokalemia (General disorders) | 3 | 3 | 1 | 1
Constipation (Gastrointestinal disorders) | 4 | 1 | 2 | 2
Dizziness (General disorders) | 2 | 3 | 1 | 1
Hypercalcemia (General disorders) | 4 | 0 | 2 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 1 | 3 | 3
Insomnia (General disorders) | 4 | 1 | 1 | 1
Hypothyroidism (General disorders) | 1 | 0 | 4 | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1 | 1
Colitis (Gastrointestinal disorders) | 3 | 2 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 1 | 4 | 4
Headache (General disorders) | 1 | 1 | 3 | 3
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 5 | 5
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 3 | 0 | 1 | 1
Leukocytosis (Blood and lymphatic system disorders) | 4 | 0 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 2 | 0 | 2 | 2
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 2
Urinary frequency (Renal and urinary disorders) | 3 | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 3 | 0 | 1 | 1
White blood cell decreased (Blood and lymphatic system disorders) | 2 | 1 | 1 | 1
Urinary tract infection (Infections and infestations) | 5 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 1 | 1 | 1
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 3 | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 2
Blood bilirubin increased (Blood and lymphatic system disorders) | 1 | 1 | 2 | 2
Ascites (Gastrointestinal disorders) | 0 | 2 | 1 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0
Hyponatremia (General disorders) | 0 | 2 | 2 | 2
Hepatobiliary disorders - Other, specify (Gastrointestinal disorders) | 1 | 0 | 2 | 2
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 1
Hypoxia (Cardiac disorders) | 3 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Allergic reaction (General disorders) | 0 | 1 | 1 | 1
Cardiac disorders - Other, specify (Cardiac disorders) | 1 | 0 | 1 | 1
Dehydration (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 2 | 0 | 0 | 0
Thromboembolic event (Blood and lymphatic system disorders) | 3 | 0 | 0 | 0
Hyperuricemia (Renal and urinary disorders) | 2 | 0 | 0 | 0
Lung infection (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Anorectal infection (Infections and infestations) | 0 | 1 | 0 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Cardiac disorders - Cardiac troponin T increased (Cardiac disorders) | 1 | 0 | 0 | 0
Gastric hemorrhage (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 1
Penile pain (General disorders) | 0 | 0 | 1 | 1
Portal vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Spermatic cord obstruction (General disorders) | 1 | 0 | 0 | 0
Stridor (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Vasovagal reaction (Nervous system disorders) | 0 | 1 | 0 | 0
Delirium (Nervous system disorders) | 1 | 0 | 0 | 0
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify* (General disorders) | 3 | 2 | 1 | 1
Encephalopathy (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Anxiety (General disorders) | 2 | 0 | 0 | 0
Blurred vision (General disorders) | 1 | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Dry mouth (General disorders) | 1 | 1 | 0 | 0
Gait disturbance (Nervous system disorders) | 2 | 0 | 0 | 0
Investigations - Other, specify (Investigations) | 0 | 1 | 1 | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1
Nervous system disorders - Other, specify (Nervous system disorders) | 1 | 0 | 1 | 1
Neutrophil count decreased (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0
Pelvic pain (Renal and urinary disorders) | 1 | 0 | 1 | 1
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 2
Social circumstances - Other, specify (Nervous system disorders) | 1 | 0 | 1 | 1
Toothache (Nervous system disorders) | 1 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 2 | 0 | 0 | 0
Urinary tract pain (Renal and urinary disorders) | 1 | 0 | 1 | 1
Vaginal pain (General disorders) | 2 | 0 | 0 | 0
Weight gain (Metabolism and nutrition disorders) | 0 | 0 | 2 | 2
Adrenal insufficiency (General disorders) | 1 | 0 | 0 | 0
Hyperhidrosis (Nervous system disorders) | 1 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 1 | 0 | 0 | 0
Uveitis (General disorders) | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-02-14): https://cdn.clinicaltrials.gov/large-docs/43/NCT04021043/Prot_SAP_001.pdf
  • Informed Consent Form (2020-04-15): https://cdn.clinicaltrials.gov/large-docs/43/NCT04021043/ICF_000.pdf